CLINICAL TRIAL: NCT07343817
Title: Ultrasonic Evaluation of Metoclopramide With or Without Dexamethasone on Gastric Motility in Traumatic Patients
Brief Title: IV Injection of Metoclopramide With or Without Dexamethasone
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ahmed Nassar Ibrahim Mohammed (Other)
Collaborators: Assiut University (Other)
Responsible Party: Sponsor-Investigator, Ahmed Nassar Ibrahim Mohammed, Resident doctor, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Anesthesia Department
Record Dates: First submitted 2025-12-15; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Trauma Injury
Keywords: Poly trauma
MeSH Terms: conditions — Accidental Injuries | interventions — Dexamethasone; Metoclopramide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (2):
- Metoclopramide (Experimental): Drug used to assessment
  Interventions: Combination Product: Dexamethasone; Diagnostic Test: Ultrasonography assessment
- Dexamethasone (Experimental): Drug used to assessment
  Interventions: Combination Product: Dexamethasone; Diagnostic Test: Ultrasonography assessment

INTERVENTIONS:
Combination Product: Dexamethasone — IV infection
  Other Names: Metoclopramide
Diagnostic Test: Ultrasonography assessment — Assessment of gastric motility by ultrasonography

SUMMARY:
Reflux and the aspiration of gastric contents have always been important focal points. Previous study stated that trauma is an important factor in aspiration pneumonia.

Often, emergency trauma patients have residual gastric contents due to the ingestion of food before injury, the accidental swallowing of nasal and/or oral blood after injury, and delayed gastric emptying due to stress, pain, or the use of opioids.

During sedation or general anesthesia, such satiated patients are often at risk of aspiration due to a reduction in lower esophageal sphincter tension and the protective inhibition of the airway reflex.

Perioperative gastric ultrasound can be performed at a bedside ultrasound unit; it can safely, non-invasively, conveniently, and effectively evaluate the fullness of a patient's stomach and the nature of their gastric contents.

It can also be used in the selection of an appropriate method for the anesthetic induction process and can reduce the risk of vomiting, aspiration, and related complications.

As a gastric motility-promoting drug, metoclopramide can accelerate gastric emptying.

Dexamethasone reduced the incidence of nausea and vomiting and improve gastric motility.

DETAILED DESCRIPTION:
PATIENTS AND METHODS Study design / Prospective randomized controlled trial study sitting/this study will be conducted in Assiut University Trauma Center Hospital.

Patients will be randomly allocated into two groups:

* Group (1) : intravenous infusion of metoclopramide 8mg
* Group (2) : intravenous infusion of metoclopramide 8mg with infusion of dexamethasone 8mg INCLUSION CRITERIA

  1. Traumatic patients undergo emergency operations
  2. 18-60 years of age
  3. 155-180 cm in height
  4. Body mass index <30 kg/m2 EXCLUSION CRITERIA

  <!-- -->

  1. A history of diseases of important organs, such as diabetes, gastro-paresis, liver and kidney dysfunction, and cardiopulmonary insufficiency.
  2. Contraindications for metoclopramide or dexamethasone treatment.
  3. Taking opioids or drugs that affect gastric motility.
  4. A history of esophageal, gastric, or upper abdominal surgery.
  5. A need for immediate emergency surgery, resulting in insufficient study time (120 min).
  6. Inability of the patient or their family to understand the study protocol.

TECHNICAL PROCEDURES

All patients who will be admitted to Assiut University Trauma Center Hospital included in this study will be connected to non-invasive blood pressure, ECG, and pulse oximetry then divided into two groups:

Group (1): Receive intravenous infusion of metoclopramide 8mg Group (2): Receive intravenous infusion of metoclopramide 8mg with infusion of dexamethasone 8mg Then these patients will be examined by ultrasound (S-Nerve Series, Sono Co., Ltd., China, fitted with a 3-5 MHz convex array probe).

The probe will be placed in the sagittal position under the xiphoid process next to the upper abdomen, and the abdominal imaging mode will be selected.

The left lobe of the liver and the abdominal aorta are anatomical marks on the section of the ultrasound image.

First, the patient will be placed in a supine position and undergo a qualitative evaluation of the gastric antrum (to determine gastric contents, i.e., liquids and solids).

Then, the cross sectional area (CSA) of the gastric antrum will be measured during the interval of gastric peristalsis.

The measurement range will be from the sub-serosa to the serosa, and the average value of three measurements will be taken as the result.

Then the patient will be placed in a half-sitting/half-lying position (the head of the bed will be raised by 45°.

These steps will be repeated, and the inspection time will be limited to 5 min. All patients who met the inclusion and exclusion criteria will be fasted (food and liquids) before the procedure and won't receive any opioids or medications that might affect gastrointestinal motility.

ELIGIBILITY:
Inclusion Criteria

* Traumatic patients undergo emergency operations
* 18-60 years of age
* 155-180 cm in height
* Body mass index <30 kg/m2

Exclusion Criteria:

* A history of diseases of important organs, such as diabetes, gastro-paresis, liver and kidney dysfunction, and cardiopulmonary insufficiency.
* Contraindications for metoclopramide or dexamethasone treatment.
* Taking opioids or drugs that affect gastric motility.
* A history of esophageal, gastric, or upper abdominal surgery.
* A need for immediate emergency surgery, resulting in insufficient study time (120 min).
* Inability of the patient or their family to understand the study protocol.

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of gastric weight/volume kg/m^2 measured by ultrasonography in traumatic patients. | 2 years
  Assessment of gastric weight/volume kg/m^2 by grams measured by ultrasonography in traumatic patients.

IPD SHARING:
Plan to Share IPD: No